CLINICAL TRIAL: NCT06629779
Title: A PHASE 3, RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED STUDY OF PF-06821497 (MEVROMETOSTAT) WITH ENZALUTAMIDE IN METASTATIC CASTRATION RESISTANT PROSTATE CANCER (MEVPRO-2)
Brief Title: A Study to Learn How PF-06821497 (Mevrometostat) Works in Men With Metastatic Castration-resistant Prostate Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2321003; 2024-511652-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-09-10; First posted 2024-10-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: MEVROMETOSTAT; METASTATIC CASTRATION RESISTANT PROSTATE CANCER; PF-06821497; EZH2; enhancer of zeste homologue-2; enzalutamide; mCRPC; Prostrate Cancer; castrate resistant prostate cancer; prostatecancer-study.com; efficacy; safety; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — PF06821497; enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants will receive PF-06821497 or matching placebo in a blinded fashion, as indicated in Section 6.1. Participants, investigators and site staff, and sponsor staff will be aware that participants in both study arms are receiving enzalutamide. Enzalutamide will be provided in an open-label manner to participants in each treatment arm.
  Participants and their caregivers will be blinded to their assigned study intervention.
  Investigators and other site staff will be blinded to participants' assigned study intervention Sponsor staff will be blinded to participants' assigned study intervention, except for sponsor staff involved in the assignment or distribution of study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive PF-06821497 (875 mg) BID (twice daily) + enzalutamide 160 mg QD (once daily)
  Interventions: Drug: PF-06821497; Drug: Enzalutamide
- Arm B (Active Comparator): Participants will receive Placebo BID (twice daily) + enzalutamide 160 mg QD (once daily)
  Interventions: Drug: Placebo; Drug: Enzalutamide

INTERVENTIONS:
Drug: PF-06821497 — Oral continuous
  Other Names: Mevrometostat
  Arms: Arm A
Drug: Placebo — Oral continuous
  Arms: Arm B
Drug: Enzalutamide — Oral continuous
  Other Names: Xtandi

SUMMARY:
This study will explore whether a combination of the investigational drug PF-06821497 and enzalutamide will work better than taking enzalutamide alone in participants with mCRPC who are ARSi or abiraterone naïve.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized Phase 3 study evaluating PF-06821497 (mevrometostat) in combination with enzalutamide versus placebo in combination with enzalutamide in participants with mCRPC where no systemic anti-cancer treatments have been initiated after documentation of mCRPC with the exception of ADT (androgen deprivation therapy) and first-generation anti-androgen agents. Prior treatment with any of the ARSi's enzalutamide, darolutamide, apalutamide, or abiraterone acetate, is not permitted in any setting. Chemotherapy is permitted in the castrate sensitive setting.

This study consists of a Screening Phase, Randomization, Treatment Phase, Safety Follow-up, and Long-Term Follow-up. Participants will be randomized on a 1:1 basis to receive (Arm A) PF-06821497 in combination with enzalutamide, or (Arm B) placebo in combination with enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features.
* Metastatic disease in bone documented on bone scan, or in soft tissue documented on CT/MRI scan.
* Progressive disease in the setting of medical or surgical castration.
* ECOG performance status 0 or 1, with a life expectancy of ≥12 months as assessed by the investigator.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that make the participant inappropriate for the study.
* Known history of active inflammatory gastrointestinal disease, chronic diarrhea, or previous gastric resection or lap-band surgery.
* Clinically significant cardiovascular disease.
* Known or suspected brain metastasis or active leptomeningeal disease or clinically significant history of seizure.
* Any history of myelodysplastic syndrome, acute myeloid leukemia, or any other prior malignancy with a few exceptions.
* Participants must be treatment naïve at the mCRPC stage, eg, no cytotoxic chemotherapy, radio-ligand therapy (i.e. 177Lu- PSMA-617), CDK4/6 inhibitors, 5-alpha reductase inhibitors for prostate cancer in any setting, androgen receptor signaling inhibitors (ARSi) including enzalutamide, apalutamide, darolutamide, poly ADP-ribose polymerase (PARP) monotherapy or other systemic anti-cancer treatment with the following exceptions:

  1. Treatment with first-generation antiandrogen (ADT) agents;
  2. Docetaxel treatment is allowed for mCSPC, as long as no signs of failure, or disease progression occurred during treatment or within 3 months of treatment completion.
* Previous administration with an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention (whichever is longer).
* Inadequate organ function.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 900 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | Randomization up to approximately 3 years
  rPFS is defined as the time from the date of randomization to first objective evidence of radiographic progression as assessed in soft tissue per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or in bone per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) guidelines by BICR, or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Randomization up to approximately 5 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
To demonstrate that PF-06821497 in combination with enzalutamide is superior to placebo in combination with enzalutamide in prolonging TTPP | Randomization up to approximately 3 years
  TTPP (alpha protected): assessed using time to first ≥2-point increase from baseline score on BPI-SF Item 3 (Worst Pain) observed at 2 consecutive visits or the initiation of short- or long-acting opioid use for pain
Duration of Response (DoR) in measurable soft tissue disease | Randomization up to approximately 3 years.
  The DoR is defined as the time from the first objective evidence of soft tissue response (CR or PR, whichever is earlier) to radiographic progression or death due to any cause whichever occurs first.
Time to prostate specific antigen (PSA) progression. | Randomization up to approximately 3 years
  Time from the date of randomization to the date of the first PSA progression. PSA progression is defined as a ≥25% increase in PSA with an absolute increase of ≥2 ng/mL above the nadir (or baseline for participants with no PSA decline), confirmed by a second consecutive PSA value at least 21 days later.
Prostate Specific Antigen Response | Randomization up to approximately 3 years.
  Proportion of participants with PSA response ≥50% in participants with detectable PSA values at baseline.
Time to initiation of antineoplastic therapy. | Randomization up to approximately 3 years.
  Time from randomization to first use of new antineoplastic therapy.
Time to initiation of cytotoxic chemotherapy. | Randomization up to approximately 3 years
  Time from randomization to first use of new cytotoxic chemotherapy.
Time to first symptomatic skeletal event | Randomization up to approximately 3 years.
  Time from randomization to first symptomatic skeletal event (symptomatic bone fractures, spinal cord compression, surgery or radiation to the bone whichever is first).
Progression free survival on next line of therapy | Randomization up to approximately 3 years
  the time from the date of randomization to the first occurrence of investigator-determined disease progression (PSA progression, progression on imaging, or clinical progression) or death due to any cause, whichever occurs first, while the participant was receiving first subsequent therapy for prostate cancer.
Incidence of Adverse Events | Randomization up to approximately 5 years
  Type, incidence, severity [as graded by National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v5.0], seriousness and relationship to study medications of AEs.
To assess circulating tumor DNA (ctDNA) at baseline and on treatment to evaluate tumor burden. | Baseline up to approximately 3 years.
  Evaluation of ctDNA burden at baseline and on study.
To evaluate the PK of PF-06821497 when dosed with enzalutamide | Cycle 1 Day 15 to last PK draw at Cycle 6 Day 1 (cycle length is 28 days)
  PK characterized by pre-dose trough and post-dose plasma concentrations of PF-06821497 at selected visits
Change from baseline in patient reported pain symptoms per Brief Pain Inventory-Short Form (BPI-SF) | Randomization up to approximately 5 years
  Analysis of Brief Pain Inventory-Short Form (BPI-SF) will be based on the pain severity score (mean of individual BPI-SF items 3, 4, 5 and 6), the pain interference score (mean of items 9A-9G), and the single BPI-SF Item 3 which asks the patient to rate pain at its worst in the last 24 hours.
Change from baseline in BPI-SF Item 3 (Worst Pain) at Cycle 7 Day 1 (Week 25) | Randomization up to Week 25
  Analysis of Brief Pain Inventory-Short Form (BPI-SF) will be based on the pain severity score (mean of individual BPI-SF items 3, 4, 5 and 6), the pain interference score (mean of items 9A-9G), and the single BPI-SF Item 3 which asks the patient to rate pain at its worst in the last 24 hours.
Change from baseline in health-related quality of life (HRQoL) per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 5 years
  Change from baseline in HRQoL (FACT-P total score) will be presented. The FACT-P total score will be calculated based on the participant responses to the 39 items in the FACT-P questionnaire. Each item is rated on a 0 to 4 Likert-type scale and then combined to produce the FACT-P total score (0-156), with higher scores representing better health-related quality of life.
Change from baseline in patient reported health status per European Quality of Life 5-Dimension 5 Level (EQ-5D-5L) | Randomization up to approximately 5 years
  Participants will self-rate their current state of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression by choosing 1 of 5 possible responses that record the level of severity (no problems, slight problems, moderate problems, severe problems, or extreme problems) within each dimension. The questionnaire also includes a visual analog scale to self-rate general health state on a scale from "the worst health you can imagine" to "the best health you can imagine."
Symptomatic toxicity as measured by items from the Patient-Reported Outcome CTCAE (PRO-CTCAE) | Randomization up to approximately 5 years
  Each selected PRO-CTCAE items will be assessed related to one or more attributes that include counts for the frequency, severity, and/or interference with usual or daily activities.
Time to definitive deterioration in patient-reported health related quality of life (HRQoL) per FACT-P | Randomization up to approximately 5 years
  Defined as the time from randomization to onset of definitive deterioration in FACT-P total score, which is defined as >10 point decrease from baseline and no subsequent observations with a <10 point decrease from baseline FACT-P total score

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (238):
- United States (40):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Goodyear, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - Highlands Oncology, Fayetteville, Arkansas
  - Arkansas Urology - Little Rock, Little Rock, Arkansas
  - Highlands Oncology, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Los Angeles Cancer Network (LACN), Anaheim, California
  - Los Angeles Cancer Network (LACN), Fountain Valley, California
  - Los Angeles Cancer Network (LACN), Glendale, California
  - Los Angeles Cancer Network (LACN), Los Angeles, California
  - Medical Oncology Associates of San Diego, San Diego, California
  - Accellacare of Duly, Lisle, Illinois
  - Duly Health and Care (Bone Scintigraphy), Lisle, Illinois
  - Blessing Hospital, Quincy, Illinois
  - Blessing Physician Services, Quincy, Illinois
  - Duly Health and Care (CT and MRI), Westmont, Illinois
  - Adult & Pediatric Urology, PC, Omaha, Nebraska
  - CHRISTUS St. Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Montefiore Medical Center - Medical Park, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Salisbury VA Medical Center, Salisbury, North Carolina
  - AUC Urologists, LLC, Myrtle Beach, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - USA Clinical Trials, San Antonio, Texas
  - Northwest Medical Specialties, PLLC, Bonney Lake, Washington
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - Harborview Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Argentina (9):
  - Centro de Urología (CDU), CABA, Buenos Aires
  - Hospital Sirio Libanes, Capital Federal, Buenos Aires
  - Imagenes Mdq, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro Medico Privado CEMAIC, Capital, Córdoba Province
  - Hospital Privado Universitario de Córdoba, Córdoba, Córdoba Province
  - IMAXE, Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - Centro Medico Fleischer, Buenos Aires
- Brazil (18):
  - Oncocentro Servico Medicos e Hospitalares Ltda, Fortaleza, Ceará
  - Hospital São Carlos, Fortaleza, Ceará
  - Oncocentro Oncologia, Fortaleza, Ceará
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador, Estado de Bahia
  - Hospital Da Bahia, Salvador, Estado de Bahia
  - Clinica Amo - Rio Vermelho, Salvador, Estado de Bahia
  - Hospital Sirio Libanes, Brasília, Federal District
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - MedPlex Eixo Norte, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova AD, Gabrovo
  - "University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski" EAD, Pleven
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sofiamed, Sofia
  - Complex Oncology Center Stara Zagora EOOD, Stara Zagora
- Canada (6):
  - Prostate Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Lakeridge Health, Oshawa, Ontario
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- Chile (10):
  - IC La Serena Research, La Serena, Coquimbo Region
  - Clinica Universidad Catolica del Maule, Talca, Maule Region
  - Centro de Investigacion Clinica del Sur, Temuco, Región de la Araucanía
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Fundación Arturo López Pérez, Providencia, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez, Providencia, Santiago Metropolitan
  - Oncovida, Providencia, Santiago Metropolitan
  - Centro de Estudios Clínicos SAGA, Santiago, Santiago Metropolitan
  - FALP, Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (29):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University School of Medicine, Shantou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People' Hospital, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang/nanhu
  - Peking University Third Hospital, Beijing
  - First Affiliated Hospital of China Medical University, Shenyang
- Czechia (8):
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Fakultní nemocnice Ostrava, Ostrava - Poruba, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Multiscan, Pardubice, Pardubický kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha 10
  - Urocentrum Praha, Prague, Praha 2
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Krajská nemocnice Liberec, Liberec
- Denmark (3):
  - Næstved Sygehus, Næstved, Region Sjælland
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Vejle Sygehus, Vejle, Region Syddanmark
- Finland (5):
  - Oulun yliopistollinen sairaala, Oulu, North Ostrobothnia
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki university hospital, Helsinki
- France (11):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Leon Berard, Lyon Cedex08, Auvergne-Rhône-Alpes
  - Hopitaux Universitaire de Strasbourg - Hopital Hautepierre, Strasbourg, Bas-rhin
  - CHRU de Brest, Brest, Finistère
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire, Ille-et-vilaine
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - Institut Jean Godinot, Reims, Marne
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand
  - Institut Godinot, Reims
- Germany (4):
  - Studienpraxis Urologie, Nürtingen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (5):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Alexandra General Hospital of Athens, Athens, Attikí
  - Athens Medical Center, Athens, Attikí
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
  - University General Hospital of Larissa, Larissa, Thessalía
- Hungary (4):
  - Borsod-Abaúj-Zemplén Vármegyei Központi Kórház és Egyetemi Oktatókórház, Miskolc, Borsod-Abauj Zemplen county
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Nograd Varmegyei Szent Lazar Korhaz, Salgótarján, Nógrád megye
  - Országos Onkológiai Intézet, Budapest, Pest County
- Italy (10):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Ospedale San Raffaele, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Azienda Ospedaliera Santa Maria Terni, Terni
  - APSS- Presidio Ospedaliero S. Chiara, Trento
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Japan (15):
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - Keio university hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Yamagata University Hospital, Yamagata
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Frisius Medisch Centrum, Leeuwarden, Provincie Friesland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland, Schiedam, South Holland
- New Zealand (5):
  - Imed Radiology, Tauranga, Bay of Plenty
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Christchurch Hospital, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region
  - Auckland City Hospital, Auckland
- Poland (10):
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions, Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie, Koszalin, West Pomeranian Voivodeship
  - SP ZOZ Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego w Opolu, Opole
  - Provita Profamilia, Piotrkow Trybunalski, Łódź Voivodeship
- Slovakia (3):
  - CUIMED, s.r.o., Urologicka ambulancia, Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Privatna urologicka ambulancia, s.r.o., Trenčín
- South Africa (4):
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - Wilgers Oncology Centre, Pretoria, Gauteng
  - Wits Clinical Research, Soweto, Gauteng
  - TASK Eden, George, Western Cape
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-kwangyǒkshi
  - Chungnam national university hospital, Junggu, Taejǒn-kwangyǒkshi
- Spain (5):
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- Södersjukhuset, Stockholm, Stockholms LÄN [se-01], Sweden
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (7):
  - Koç Üniversitesi Hastanesi, Istanbul, İ̇stanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul, İ̇stanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul, İ̇stanbul
  - I.E.U. Medical Point Hastanesi, Izmir, İ̇zmir
  - Sbü Gülhane Eğitim Ve Araştirma Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara University Health Practice and Research Hospitals, Ankara
- United Kingdom (5):
  - Royal Blackburn Hospital, Blackburn, Blackburn WITH Darwen
  - Mid and South Essex NHS Foundation Trust, Chelmsford, Essex
  - Royal Derby Hospital, Derby
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321003
- See also: www.mevpro2.com — https://www.pfizerclinicaltrials.com/nct06629779-metastatic-prostate-cancer-trial